CLINICAL TRIAL: NCT05072600
Title: A Pilot Study of Pembrolizumab Monotherapy as Maintenance Therapy in MIBC Patients Who Received Bladder-Preserving Trimodally Therapy and Achieved CR
Brief Title: Pembrolizumab Monotherapy Following Tri-modality Treatment for Selected Patients With Muscle-invasive Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Zhisong HE, Director of Department of Urology, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-305
Record Dates: First submitted 2021-09-18; First posted 2021-10-11 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Bladder Cancer; Bladder Neoplasms; Bladder Tumors; Urinary Bladder Cancer; Neoplasms, Bladder
Keywords: bladder cancer; radiotherapy; Pembrolizumab; tri-modality therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arm 1 (Experimental): All participants will receive pembrolizumab monotherapy per 21 days no longer than 17 cycles until disease progression or death.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab 200 mg Q3W
  Other Names: PD-1 inhibitor

SUMMARY:
This is a Phase II, single-arm, study of pembrolizumab as maintenance therapy in muscle-invasive bladder cancer (MIBC) participants who have received maximum TURBT and tri-modality treatment (TMT) and achieved CR. All participants will receive pembrolizumab monotherapy per 21 days no longer than 17 cycles until disease progression or death.

DETAILED DESCRIPTION:
Radical cystectomy (RC) has long been the standard of care for the treatment of muscle-invasive bladder cancer (MIBC). Modern RC series have demonstrated 5-yr overall survival (OS) rates of 56-66%. There has been an increasing trend of utilizing organ-preserving therapies in the management of bladder cancer over the past several decades. A multidisciplinary approach has led to the development of bladder-sparing approaches using maximal transurethral resection (TURBT) followed by radiotherapy with concomitant radio-sensitizing chemotherapy for MIBC. Multiple tri-modality treatment (TMT) series have suggested that TMT can yield favorable results in well-selected patients. The 5-yr OS is 48-75%, and 75-80% of the survivors have preserved their native bladder. Even if local recurrence occurred after concurrent radio-chemotherapy, salvage cystectomy can also bring 50-57.6% of 5-year disease-specific survival (DSS) without more complications associated with surgery. So, NCCN guidelines have regarded this TMT strategy as a preferred choice for patients with MIBC since 2019.

However, distant metastasis after TMT was still the main concern. Giacalone NJ, et al. reported that the 5-yr distant metastasis rate was 32% in MIBC patients who received an organ-preserving strategy. Up to now, there was no consensus on adjuvant therapy after concurrent radio-chemotherapy. Some retrospective studies demonstrated that adjuvant chemotherapy had no survival benefit, and only approximately 50% of patients completed the planned adjuvant chemotherapy due to intolerable toxicities.

These years, studies on PD-(L)1 inhibitors for urothelial carcinoma showed the efficacy and safety. FDA has approved indications of pembrolizumab used as 1L (selected patients) and 2L treatment for metastatic urothelial carcinoma. Checkmate-274 has reported that adjuvant immunotherapy improved disease-free survival (DFS) in MIBC patients after RC. Javelin Bladder 100 prolonged OS of mUC patients by Avelumab as maintenance therapy who achieved CR, PR or PD after 1L chemotherapy. These results support our hypothesis that, for those MIBC patients who have received bladder-preserving TMT and achieved CR, pembrolizumab monotherapy as maintenance therapy is superior to observation.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent.
2. Based on AJCC 8th edition: stage cT2-4N0M0，Urothelial carcinoma >50% and

   * Requires definitive local therapy
   * Has received maximum TURBT followed by tri-modality therapy
   * Achieved CR after tri-modality therapy, the acceptable duration of time between completion of TMT and assessment of CR was 28-90 days.
3. Tumor was located at one side of bladder wall.
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Have adequate organ function prior to the start of study intervention.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Patients judged not to be candidates for radical cystectomy; patients with pN+ or T4b disease are considered to have unresectable disease; Has any distant metastases.
4. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.
5. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
6. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
8. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
9. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a known history of Human Immunodeficiency Virus (HIV) infection.
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
19. Has had an allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-12-07 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | three years
  PFS is defined as the time from first dose of pembrolizumab to any of the following events: recurrent MIBC, nodal or distant metastases or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Song He, MD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China